CLINICAL TRIAL: NCT06943573
Title: Psilocybin-Assisted Therapy for Treatment-Resistant Depression in Bipolar II Disorder: A Randomized Controlled Trial
Brief Title: Psilocybin-Assisted Therapy for Treatment-Resistant Depression in Bipolar II Disorder
Acronym: PAT-BD-01
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lakshmi N Yatham (Other)
Responsible Party: Sponsor-Investigator, Lakshmi N Yatham, Professor, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H25-00074
Record Dates: First submitted 2025-04-01; First posted 2025-04-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Bipolar II Depression
Keywords: Bipolar Disorder; Mood Disorder; Psychedelic-assisted therapy; Psychedelics; Treatment resistant; Psilocybin; Depression
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Depression | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Double-blind, Active Placebo controlled, Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study Therapist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): 25 mg psilocybin.
  Interventions: Drug: psilocybin (25 mg)
- Placebo (Placebo Comparator): 1 mg psilocybin (micro-dose)
  Interventions: Drug: psilocybin 1mg micro-dose

INTERVENTIONS:
Drug: psilocybin (25 mg) — Single-dose psilocybin (25 mg)-assisted therapy (PAT)
  Arms: Active
Drug: psilocybin 1mg micro-dose — Single dose active placebo psilocybin-assisted therapy
  Arms: Placebo

SUMMARY:
This study is a 12-week (in addition to up to 30 days of screening) randomized, double-blind, placebo-controlled, parallel-group trial. The primary objective of this study is to assess the effectiveness, safety, and tolerability of single-dose psilocybin (25 mg)-assisted therapy in comparison to active placebo (1 mg micro-dose) psilocybin-assisted therapy in patients with bipolar II depression who have not responded to adequate trials with at least two first or second-line treatments for bipolar II depression (i.e. quetiapine, lithium, lamotrigine, sertraline, or venlafaxine as monotherapy or adjunctive therapy, or bupropion adjunctive therapy). The active placebo is a substance that looks identical to the study medication but contains less therapeutic ingredients, and thus is less capable of producing the transformative and meaningful aspects of psychedelic experience compared to the 25 mg dose. Participants will have a total of 11 study visits over a period of up to 16 weeks, which includes 5 therapy sessions from trained study therapists.

DETAILED DESCRIPTION:
Bipolar disorders (BD) are lifelong conditions characterized by recurrent episodes of depression and (hypo)mania. Statistics Canada data indicate over a million Canadians are affected by this illness. Bipolar II disorder is characterised by recurrent episodes of hypomania and depression and individuals with BD-II are symptomatic about 50% of the time despite treatment. The majority of this time is spent being depressed thus there is an urgent need to develop new treatments that are safe and effective. Psilocybin, a naturally occurring psychedelic compound found in mushrooms, has been noted to result in an increase in psychological well-being in healthy volunteers as well as have antidepressant effects when administered in conjunction with psychological support. Two recent open-label pilot trials of Psilocybin-Assisted Therapy (PAT) in treatment-resistant depression, including BD-II participants, demonstrated high response rates and excellent tolerability, thereby providing strong justification for the current study.

ELIGIBILITY:
Inclusion Criteria:

1. You are male or female aged 19 to 65 years inclusive.
2. You have a diagnosis of bipolar disorder type II, and are currently in a major depressive episode.
3. You are willing, for the entire duration of the study, to practice highly effective methods of contraception (e.g., contraceptive pills, intrauterine device or system, vasectomy and tubal ligation, or double-barrier methods of contraception) OR agree to completely abstain from heterosexual intercourse. Females who do not have childbearing potential are required to be postmenopausal for at least 1 year before the screening visit (confirmed by an FSH test) OR surgically sterile.
4. You have sufficient English language skills to understand, consent to, and comply with study requirements, study visits, and to return to the clinic for follow-up evaluations.
5. Your current medications have been at a stable dose for two weeks prior to the dosing visit.

Exclusion Criteria:

1. You have a history of psychotic symptoms.
2. You have a history of seizures.
3. You have a current unstable or inadequately treated medical illness, especially cardiovascular illness, except for the current depression.
4. You recently (i.e., within the past 6 weeks) started taking treatment for your acute bipolar depressive episode.
5. You recently (i.e., within the past 8 weeks) began structured psychotherapy (e.g., cognitive-behavioral therapy, interpersonal psychotherapy, family-focused therapy, or interpersonal and social rhythm therapy).
6. You have a history of nonresponse or intolerance to psilocybin.
7. You have, in the past 6 months, used any psychedelic drugs, including ketamine, LSD, or psilocybin-containing mushrooms.
8. You have a history of non-response to electroconvulsive therapy.
9. You are pregnant or lactating.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | Baseline to Week 3
  The Montgomery Asberg Depression Rating Scale (MADRS) will be used to measure change in depressive symptoms. Scores range from 0 to 60, and lower scores reflect better clinical outcomes.

SECONDARY OUTCOMES:
Response Rates | Week 3, Week 6, Week 12
  Patients showing ≥50% reduction in the Montgomery Asberg Depression Rating Scale (MADRS) scores from Baseline. Scores range from 0 to 60, and lower scores reflect better clinical outcomes.
Remission Rates | Endpoint
  Defined as Montgomery Asberg Depression Rating Scale (MADRS) scores ≤ 10 and Young Mania Rating Scale (YMRS) scores ≤ 8. Scores for the MADRS range from 0 to 60, with lower scores reflecting better clinical outcomes. Scores for the YMRS range from 0 to 60, with lower scores reflecting better clinical outcomes.
Treatment-emergent manic/hypomanic events | 12 weeks
  The Young Mania Rating Scale (YMRS) will be used to determine the presence of any treatment-emergent manic or hypomanic events from baseline to endpoint. Scores range from 0 to 60, and lower scores reflect better clinical outcome
Mean change in depressive symptoms | Week 6 and 12
  The Montgomery Asberg Depression Rating Scale (MADRS) will be used to measure mean change in depressive symptoms. Scores range from 0 to 60, and lower scores reflect better clinical outcomes.
Subjective depressive symptoms | 12 weeks
  The Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR) will be used to measure change in subjective depressive symptoms from baseline to endpoint. Scores on the QIDS-SR range from 0 to 27; lower scores on the QIDS-SR reflect better clinical outcomes.
Symptoms of anhedonia | 12 weeks
  The Snaith-Hamilton Pleasure Scale (SHAPS) will be used to measure change in subjective symptoms of anhedonia from baseline to endpoint. Scores on the SHAPS range from 0 to 42; higher SHAPS scores indicate a reduced ability to experience pleasure and reduced capacity to feel pleasure.
Objective anxiety symptoms | 12 weeks
  The Hamilton Anxiety Rating Scale (HAM-A) will be used to measure change in objective anxiety symptoms from baseline to endpoint. Scores range from 0 to 56 and lower scores reflect better clinical outcomes.
Overall psychiatric status | 12 weeks
  The Clinical Global Impression - severity & change scales will be used to measure change in global severity and global improvement in symptoms from baseline to endpoint. Scores range from 3 to 42, and higher scores reflect worsening in overall psychiatric status.
Psychotic symptoms | 12 weeks
  The Positive and Negative Syndrome Scale (PANSS) will be used to measure change in psychotic symptoms from baseline to endpoint. Scores range from 7 to 49, and lower scores reflect better clinical outcomes.
Subjective cognitive functioning | 12 weeks
  The Cognitive Complaints in Bipolar Disorder Risk Assessment (COBRA) scale will be used to measure change in subjective cognitive functioning from baseline to endpoint. COBRA scores range from 0 to 48, and lower scores reflect better outcomes.
Objective cognitive functioning | 12 weeks
  The Screen for Cognitive Impairment in Psychiatry (SCIP) will be used to measure change in objective cognitive functioning from baseline to endpoint. Higher scores reflect better outcomes.
Sleep quality | 12 weeks
  The Pittsburgh Sleep Quality Index (PSQI) will be used to measure changes in sleep quality and disturbance from baseline to endpoint. Lower scores reflect better sleep quality.
Quality of Life assessed by QoL.BD | 12 weeks
  The Brief Quality of Life in Bipolar Disorder (QoL.BD) will be used to measure change in quality of life from baseline to endpoint. Higher scores reflect higher quality of life.
Daily functioning | 12 weeks
  The Functioning Assessment Short Test (FAST) will be used to measure change in daily functioning from baseline to endpoint. Scores range from 0 to 72 with lower scores reflecting better daily functioning.
Suicidal thoughts and behaviours | 12 weeks
  The Columbia-Suicide Severity Rating Scale (C-SSRS) will be used to measure change in suicidal thoughts and behaviours from baseline to endpoint. Scores range from 0 to 37, and lower scores reflect better clinical outcomes.
MEQ30 | Dosing Visit (Day 0)
  Psychedelic experience will be measured by the MEQ30. Scores range from 30 to 150; higher scores reflect stronger (more profound) experiences.
Clinician's perspective on the therapeutic relationship | Baseline and Week 1
  The Therapeutic Relationship will be measured with the Scale to Assess the Therapeutic Relationship - Clinician version (STAR-C). Scores range from 0 to 48 respectively; higher scores reflect better therapeutic relationships.
Patient's perspective on the therapeutic relationship | Baseline and Week 1
  The Therapeutic Relationship will be measured with the Scale to Assess the Therapeutic Relationship - Patient version (STAR-P). Scores range from 0 to 48 respectively; higher scores reflect better therapeutic relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Lakshmi N Yatham, Principal Investigator — UBC Department of Psychiatry
Locations (3):
- Canada (3):
  - Djavad Mowafaghian Centre for Brain Health, Vancouver, British Columbia
  - Department of Psychiatry, University of Ottawa, The Ottawa Hospital, Ottawa, Ontario
  - Department of Psychiatry, University of Toronto, University Health Network,, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No